CLINICAL TRIAL: NCT03715452
Title: Minimizing Radiographic Contrast Administration During Coronary Angiography Using a Novel Contrast Reduction System: A Multicenter Observational Study of the DyeVert™ Plus Contrast Reduction System
Brief Title: DyeVert™ Plus Contrast Reduction System Multicenter Observational Study
Status: Completed | Type: Observational
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-6579
Record Dates: First submitted 2018-10-15; First posted 2018-10-23 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- DyeVert Plus Contrast Reduction System: DyeVert Plus Contrast Reduction System
  Interventions: Device: DyeVert Plus Contrast Reduction System

INTERVENTIONS:
Device: DyeVert Plus Contrast Reduction System — The DyeVert Plus System interfaces with standard manifold systems to provide real-time contrast monitoring and reduce the amount of contrast used in catheterization procedures while maintaining fluoroscopic image quality. System components include a disposable, single-use, sterile DyeVert Plus Disposable Kit that contains a Smart Syringe and DyeVert Plus Module, which is connected to a standard manifold and provides fluid pathway resistance modulation via a dedicated diversion valve. The diversion valve self-adjusts to the manual injection pressure to divert some of the contrast media into the reservoir chamber within the module. This diverted volume of contrast media does not enter the patient.

SUMMARY:
This is a prospective, single arm, multi-center, observational clinical study of the DyeVert Plus System. The DyeVert Plus System is an FDA-cleared device designed to reduce contrast media volume delivered during angiography and permit real-time contrast media volume monitoring.

DETAILED DESCRIPTION:
The purpose of this observational study is to evaluate the amount of contrast media saved using DyeVert Plus in coronary angiographic and/or interventional procedures performed with manual injection and evaluate the impact of predetermined thresholds and real-time monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo CAG and/or PCI
* Baseline estimated glomerular filtration rate (eGFR) of ≥20 and ≤60 mL/ min/1.73 m2

Exclusion Criteria:

* Acute ST-elevation myocardial infarction or known coronary artery fistulas
* Body mass index (BMI) >40
* Currently pregnant
* Undergoing a chronic total occlusion procedure or optical coherence tomography analysis
* Planning to undergo transcatheter aortic valve replacement within 72 hr of the index procedure
* A condition known to require large volumes of contrast (>10 mL) for each injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects undergoing diagnostic coronary angiography (CAG) and/or percutaneous coronary interventional (PCI) procedures performed with manual injections
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Harbor UCLA Medical Center, Torrance, California
  - Atlanta VA Medical Center, Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - WakeMed Heart and Vascular, Raleigh, North Carolina
  - Christ Hospital, Heart and Vascular Center, Lindner Research Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DyeVert™ Plus Contrast Reduction System: DyeVert Plus Contrast Reduction System
  The DyeVert Plus System interfaces with standard manifold systems to provide real-time contrast monitoring and reduce the amount of contrast used in catheterization procedures while maintaining fluoroscopic image quality. System components include a disposable, single-use, sterile DyeVert Plus Disposable Kit that contains a Smart Syringe and DyeVert Plus Module, which is connected to a standard manifold and provides fluid pathway resistance modulation via a dedicated diversion valve. The diversion valve self-adjusts to the manual injection pressure to divert some of the contrast media into the reservoir chamber within the module. This diverted volume of contrast media does not enter the patient.
Period: Overall Study
Arm/Group | DyeVert™ Plus Contrast Reduction System
Started | 114
Completed | 114
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- DyeVert™ Plus Contrast Reduction System: Dyevert™ Plus Contrast Reduction System
  DyeVert Plus Contrast Reduction System: The DyeVert Plus System interfaces with standard manifold systems to provide real-time contrast monitoring and reduce the amount of contrast used in catheterization procedures while maintaining fluoroscopic image quality. System components include a disposable, single-use, sterile DyeVert Plus Disposable Kit that contains a Smart Syringe and DyeVert Plus Module, which is connected to a standard manifold and provides fluid pathway resistance modulation via a dedicated diversion valve. The diversion valve self-adjusts to the manual injection pressure to divert some of the contrast media into the reservoir chamber within the module. This diverted volume of contrast media does not enter the patient.
Arm/Group | DyeVert™ Plus Contrast Reduction System
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 86
  Race: African American | 25
  Race: Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m2] | 43 (11)
Serum creatinine (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 1.6 (0.5)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29 (5)
Comorbidities [Number; unit: participants]
  Hypertension | 110
  Coronary artery disease | 86
  Prior PCI | 60
  Diabetes | 60
  Congestive heart failure | 54
  Prior myocardial infarction | 39
  Anemia | 33
  Angina | 30
Procedure type [Count of Participants; unit: Participants]
  CAG only | 74
  CAG+PCI | 30
  PCI only | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Contrast Media Volume Saved
Description: The percentage of contrast media volume saved (diverted) over the total procedure as reported on the DyeVert Plus display at the end of each case.
Time Frame: At the time of the coronary angiography (CAG) or percutaneous coronary interventional (PCI) procedure
Measure: Mean (95% Confidence Interval); unit: % CMV savings per procedure
Arm/Group | DyeVert Plus Contrast Reduction System
Number analyzed (Participants) | 105
% CMV savings per procedure | 40.1 [38.4 to 41.8]

2. Secondary Outcome: Evaluation of Adverse Events Through Discharge (From the Index Procedure)
Description: An adverse event is defined as "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device." DyeVert Plus System-related adverse events will be collected. Additionally, contrast media-related adverse events, such as acute kidney injury and anaphylactic shock, will be collected.
Time Frame: From the time of the procedure through discharge (from the index procedure, approximately 0 - 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | DyeVert Plus Contrast Reduction System
Number analyzed (Participants) | 114
Participants | 11

ADVERSE EVENTS:
Time Frame: Procedure through discharge.
Arm/Group | DyeVert Plus Contrast Reduction System
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 11/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DyeVert Plus Contrast Reduction System (N=114)
DyeVert Plus System-Related Events (Product Issues) | 0 (0) — Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, related to the DyeVert Plus System
Acute Kidney Injury (Renal and urinary disorders) | 11 (11) — Acute kidney injury events were defined as a >0.3 mg/dL increase in serum creatinine post-procedure through discharge compared to the baseline value or through the date of, but prior to, a secondary procedure for staged procedures.
Contrast-Related Anaphylactic Shock (Immune system disorders) | 0 (0) — Based on clinical judgement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT03715452/Prot_SAP_000.pdf